CLINICAL TRIAL: NCT06858969
Title: A Phase II Clinical Study of Chidamide in Combination With PD-1 Inhibitor, Bevacizumab, and XELOX as First-Line Treatment for Metastatic Colorectal Cancer
Brief Title: Chidamide in Combination With PD-1 Inhibitor, Bevacizumab, and XELOX for Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, AIPING ZHOU, Doctor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q100
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): PD-1 inhibitor: Dose determined per the manufacturer's instructions or investigator's discretion based on patient status.
  Bevacizumab: 7.5 mg/kg via intravenous infusion every 3 weeks (Q3W).
  XELOX regimen:
  Oxaliplatin: 130 mg/m² via intravenous infusion on Day 1;
  Capecitabine: 1000 mg/m² orally twice daily on Days 1-14;
  Repeated every 3 weeks for 6 cycles.
  Maintenance therapy after 6 cycles (experimental group):
  Chidamide: Administered at the maximum tolerated dose/recommended phase II dose (MTD/RP2D), orally twice weekly (on Days 1, 4, 8, 11, 15, and 18 of each cycle), 30 minutes after meals.
  PD-1 inhibitor, Bevacizumab, and Capecitabine: Continued at the same doses and schedules as during the initial treatment phase.
  Interventions: Drug: Treatment group
- Standard-of-care control group (Active Comparator): XELOX + Bevacizumab: Doses identical to the experimental group (Oxaliplatin 130 mg/m², Capecitabine 1000 mg/m², Bevacizumab 7.5 mg/kg Q3W) for 6 cycles.
  Maintenance therapy after 6 cycles: Bevacizumab (7.5 mg/kg Q3W) and Capecitabine (1000 mg/m² orally twice daily on Days 1-14 of each cycle).
  Interventions: Drug: Standard-of-care control group

INTERVENTIONS:
Drug: Treatment group — Chidamide+XELOX + Bevacizumab+PD-1
  Arms: Treatment group
Drug: Standard-of-care control group — XELOX + Bevacizumab+PD-1
  Arms: Standard-of-care control group

SUMMARY:
This phase II, open-label, dose-escalation study aims to (1) assess the safety and tolerability of chidamide in combination with PD-1 inhibitor, bevacizumab, and XELOX as first-line therapy for treatment-naïve metastatic colorectal cancer patients, (2) establish the recommended phase II dose (RP2D) of the combination regimen, and (3) obtain preliminary efficacy data including objective response rate (ORR) and progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years, regardless of gender; Histologically confirmed unresectable metastatic/recurrent colorectal adenocarcinoma; No prior systemic antitumor therapy received for metastatic/recurrent colorectal adenocarcinoma; For subjects who have received prior neoadjuvant/adjuvant therapy, the interval between the last treatment and recurrence/progression must exceed 12 months; ECOG performance status 0-1; At least one measurable lesion (per RECIST v1.1 criteria); Expected survival ≥3 months;

Organ function must meet the following requirements prior to the first dose of the investigational drug:

1. Hematological function (no blood transfusion or growth factor administration within 14 days before screening):

   Absolute neutrophil count ≥1.5×10^9/L, Platelet count ≥100×10^9/L, Hemoglobin ≥90 g/L;
2. Hepatic and renal function (no albumin infusion within 14 days before screening):

   Total bilirubin ≤1.5×ULN, Serum albumin ≥25 g/L, ALT and AST ≤2.5×ULN (≤5.0×ULN for patients with liver metastases), Serum creatinine ≤1.5×ULN;
3. Coagulation function:

   INR ≤1.5×ULN, PT and APTT ≤1.5×ULN;
4. Urinalysis:

Urine protein <2+; for subjects with baseline urine protein ≥2+, 24-hour urine protein quantification must be <1 g; Subjects (including females and males) must agree to use effective contraception from signing the informed consent form until 180 days after the last dose of the investigational drug. Females of childbearing potential must not be pregnant or breastfeeding; Prior treatment-related adverse events (AEs) must have resolved to ≤Grade 1 (per NCI CTCAE v5.0, except alopecia); Voluntary participation in this clinical trial with written informed consent.

Exclusion Criteria:

* Subjects with known tumor microsatellite instability-high (MSI-H) status.

Prior treatment with histone deacetylase (HDAC) inhibitors, including but not limited to chidamide or entinostat.

Prior postoperative adjuvant therapy targeting EGFR or VEGF/VEGFR, including bevacizumab, cetuximab, panitumumab, aflibercept, regorafenib, or biosimilars of these agents.

Prior treatment with T-cell co-stimulation or immune checkpoint therapies, including CTLA-4 inhibitors, PD-1/PD-L1/PD-L2 inhibitors, or other T-cell-targeted drugs.

Active hepatitis B (HBV DNA ≥ 500 IU/mL) or hepatitis C (HCV antibody-positive with HCV-RNA above the lower limit of detection).

Central nervous system (CNS) metastases or leptomeningeal metastases.

History of cerebrovascular accident, myocardial infarction, unstable angina, or poorly controlled arrhythmia within the past 6 months (including QTc interval ≥ 450 ms in males or ≥ 470 ms in females, calculated via Fridericia's formula).

Clinically uncontrolled pleural effusion, ascites, or pericardial effusion requiring intervention and deemed ineligible by the investigator.

Cardiac dysfunction (NYHA class III/IV) or left ventricular ejection fraction (LVEF) < 50% on echocardiography.

History of other malignancies within 5 years prior to signing informed consent, except cured basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ.

Immunodeficiency, including HIV positivity, congenital/acquired immune deficiency, or history of organ/allogeneic bone marrow transplantation.

Active autoimmune disease or autoimmune disease history (e.g., interstitial pneumonia, colitis, hepatitis, thyroid dysfunction). Exceptions: vitiligo, childhood asthma/allergies in remission without adult intervention, stable hypothyroidism on hormone replacement, or type I diabetes on stable insulin.

Uncontrolled hypertension (systolic ≥ 150 mmHg and/or diastolic ≥ 100 mmHg).

History of hypertensive crisis or hypertensive encephalopathy.

Systemic corticosteroid use (>10 mg prednisone daily or equivalent) or immunosuppressants within 2 weeks prior to treatment.

Active systemic infection requiring IV antibiotics >7 days within 2 weeks prior to treatment.

Anti-tuberculosis therapy within 1 year prior to treatment.

History of substance abuse, alcoholism, or psychiatric/neurological disorders (e.g., epilepsy, dementia, hepatic encephalopathy).

Participation in other clinical trials with investigational drugs within 4 weeks prior to treatment.

Hypersensitivity to macromolecular protein preparations or any component of the study drugs.

Live vaccination within 4 weeks prior to treatment.

Major surgery within 4 weeks prior to treatment or planned during the study.

Hemoptysis (≥2.5 mL of bright red blood) or clinically significant gastrointestinal bleeding within 2 months prior to treatment.

Current or history of gastrointestinal obstruction, unless resolved with treatment and deemed eligible by the investigator.

Hemorrhagic tendency or clinically significant coagulopathy.

Unhealed wounds, active ulcers, or untreated fractures.

Recent use of antiplatelet/anticoagulant agents:

Aspirin (>325 mg/day) or clopidogrel (>75 mg/day) within 10 days prior to treatment;

Therapeutic anticoagulation (except low-molecular-weight heparin) within 2 weeks prior to treatment.

Gastrointestinal abnormalities affecting drug absorption (e.g., dysphagia, chronic diarrhea, gastrectomy).

Any condition that, in the investigator's judgment, increases study risk, confounds results, or renders the patient unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-04-09 (Estimated); Primary Completion 2026-01-08 (Estimated); Study Completion 2028-01-08 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  Evaluated using RECIST 1.1 criteria

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  Evaluated using RECIST 1.1 criteria
Overall Survival (OS) | 24 months
  Evaluated using RECIST 1.1 criteria
safety | 24 months
  Based on NCI-CTCAE 5.0 criteria.